CLINICAL TRIAL: NCT01937754
Title: Study of the Effects of an Oral Nitric Oxide Supplement on Functional Capacity and Blood Pressure in Healthy Adults With Prehypertension
Brief Title: Study of the Effects of an Oral Nitric Oxide Supplement on Blood Pressure in Prehypertensive Adults
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neogenis Laboratories (Other)
Responsible Party: Principal Investigator, Dr. Ernst Schwarz, Attending Cardiologist, Professor of Medicine, Neogenis Laboratories
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Neo-4085
Record Dates: First submitted 2013-08-29; First posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Prehypertension
Keywords: Prehypertension; Nitric Oxide; Blood Pressure; Functional Capacity; Quality of Life
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Nitric Oxide supplement (Active Comparator)
  Interventions: Dietary Supplement: Nitric Oxide supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nitric Oxide supplement — Lozenge consisting of beetroot and 75 mg caffeine
  Other Names: Neo40 Daily
  Arms: Nitric Oxide supplement
Dietary Supplement: Placebo — Same form factor and flavor as test lozenge but contains no active ingredients
  Arms: Placebo

SUMMARY:
Oral supplementation of Neo40(TM), a nitrate lozenge, will reduce blood pressure in healthy adults with clinical prehypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 to 80 years
* Two blood pressure readings of >/=135/80 mmHg at rest, thus representing prehypertension
* Informed consent

Exclusion Criteria:

* Existence of any significant internal or cardiovascular disease;
* Current use of any antihypertensive medication.
* Inability to give informed consent, or fill out standard questionnaires or inability to follow up clinically.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Reduction in Systolic and Diastolic Blood Pressure Readings | 30 days
  Two blood pressure readings at rest will be taken at baseline and again after thirty days during the follow-up appointment.

SECONDARY OUTCOMES:
Improvement in Functional Capacity | 30 days
  Participant will take a six minute walk test at baseline and again after thirty days during the follow-up appointment. Achieved distances will be measured and recorded.

OTHER OUTCOMES:
Improvement in Quality of Life | 30 days
  Participants will fill out a standardized quality of life questionnaire at baseline and again after thirty days during the follow-up appointment. Summary component scores will be recorded and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Schwarz, MD, PhD, Principal Investigator — California Medical Institute, Cedars Sinai Medical Center
Locations (1):
- California Medical Institute, Beverly Hills, California, United States